CLINICAL TRIAL: NCT02529046
Title: Effect of Conjugated Linoleic Acid Associated With Aerobic Exercise on Body Fat and Lipid Profile in Obese Women: A Randomized, Double-blinded and Placebo-controlled Trial
Brief Title: Conjugated Linoleic Acid in Obese Women
Acronym: CLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Edilson Serpeloni Cyrino, Professor, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESCyrino
Record Dates: First submitted 2015-08-04; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Lipid Metabolism Disorders; Obesity
MeSH Terms: conditions — Lipid Metabolism Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise associated with CLA (Active Comparator): CLA group received supplementation at a dose of 3.2 g/day (mixture of isomers of CLA isomers predominantly c9, t11 - 50% and c12, t10 - 80%).
  Interventions: Dietary Supplement: CLA
- Aerobic exercise (Placebo Comparator): Placebo group received 4 g/day of olive oil.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Dietary Supplement: CLA — CLA group received supplementation at a dose of 3.2 g/day (mixture of isomers of CLA isomers predominantly c9, t11 - 50% and c12, t10 - 80%). Aerobic exercise associated with CLA
  Arms: Aerobic exercise associated with CLA
Behavioral: Placebo — Placebo group received 4 g/day of olive oil. Aerobic exercise
  Arms: Aerobic exercise

SUMMARY:
In this trial, the investigators analyzed the effects of eight weeks of CLA supplementation associated with aerobic exercise on body fat and lipid profile in obese women.

DETAILED DESCRIPTION:
The aim of this investigation was to analyze the effects of eight weeks of CLA supplementation associated with aerobic exercise on body fat and lipid profile in obese women. The investigators performed a randomized, double-blinded and placebo-controlled trial with 28 obese women who received 3.2 g/d of CLA or 4 g/d of olive oil (placebo group) while performing an 8-week protocol of aerobic exercise. Dietary intake (food record), body fat (DXA) and biochemical analysis (blood sample) were assessed before and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Had no signs or symptoms of disease
* No orthopedic injuries
* Must be inactive or moderately active (defined as performing any type of physical exercise less than twice a week)
* Must be non-smokers
* Must be free from the use of ergogenic aids
* Had no metabolic disorders or chronic degenerative diseases
* Not use drug therapy for body mass loss.

Exclusion Criteria:

* Had frequency to training sessions below 85% of the total sessions

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2007-03; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Body fat | 8 weeks
  Dual-energy X-ray absorptiometry

SECONDARY OUTCOMES:
Total cholesterol | 8 weeks
  Blood analysis
Triglycerides | 8 weeks
  Blood analysis
High-density lipoprotein | 8 weeks
  Blood analysis
Low-density lipoprotein | 8 weeks
  Estimated by Friedewald formula
Trunk fat | 8 weeks
  Dual-energy X-ray absorptiometry
Arm fat | 8 weeks
  Dual-energy X-ray absorptiometry
Leg fat | 8 weeks
  Dual-energy X-ray absorptiometry

OTHER OUTCOMES:
Body mass | 8 weeks
  Urano, model PS 180
Maximum oxygen uptake | 8 weeks
  incremental treadmill test

CONTACTS AND LOCATIONS:
Overall Officials: Edilson Cyrino, PhD, Study Chair — Universidade Estadual de Londrina
Locations (1):
- Universidade Estadual de Londrina, Londrina, Paraná, Brazil

REFERENCES:
- [Result] Adams RE, Hsueh A, Alford B, King C, Mo H, Wildman R. Conjugated linoleic Acid supplementation does not reduce visceral adipose tissue in middle-aged men engaged in a resistance-training program. J Int Soc Sports Nutr. 2006 Dec 13;3(2):28-36. doi: 10.1186/1550-2783-3-2-28. PMID 18500970
- [Result] Alkerwi A, Vernier C, Crichton GE, Sauvageot N, Shivappa N, Hebert JR. Cross-comparison of diet quality indices for predicting chronic disease risk: findings from the Observation of Cardiovascular Risk Factors in Luxembourg (ORISCAV-LUX) study. Br J Nutr. 2015 Jan 28;113(2):259-69. doi: 10.1017/S0007114514003456. Epub 2014 Dec 5. PMID 25475010
- [Result] Banu J, Bhattacharya A, Rahman M, O'Shea M, Fernandes G. Effects of conjugated linoleic acid and exercise on bone mass in young male Balb/C mice. Lipids Health Dis. 2006 Mar 23;5:7. doi: 10.1186/1476-511X-5-7. PMID 16556311
- [Result] Bhattacharya A, Banu J, Rahman M, Causey J, Fernandes G. Biological effects of conjugated linoleic acids in health and disease. J Nutr Biochem. 2006 Dec;17(12):789-810. doi: 10.1016/j.jnutbio.2006.02.009. Epub 2006 May 2. PMID 16650752
- [Result] Blankson H, Stakkestad JA, Fagertun H, Thom E, Wadstein J, Gudmundsen O. Conjugated linoleic acid reduces body fat mass in overweight and obese humans. J Nutr. 2000 Dec;130(12):2943-8. doi: 10.1093/jn/130.12.2943. PMID 11110851
- [Result] Carvalho RF, Uehara SK, Rosa G. Microencapsulated conjugated linoleic acid associated with hypocaloric diet reduces body fat in sedentary women with metabolic syndrome. Vasc Health Risk Manag. 2012;8:661-7. doi: 10.2147/VHRM.S37385. Epub 2012 Dec 13. PMID 23271912
- [Result] Colakoglu S, Colakoglu M, Taneli F, Cetinoz F, Turkmen M. Cumulative effects of conjugated linoleic acid and exercise on endurance development, body composition, serum leptin and insulin levels. J Sports Med Phys Fitness. 2006 Dec;46(4):570-7. PMID 17119522
- [Result] de Deckere EA, van Amelsvoort JM, McNeill GP, Jones P. Effects of conjugated linoleic acid (CLA) isomers on lipid levels and peroxisome proliferation in the hamster. Br J Nutr. 1999 Oct;82(4):309-17. PMID 10655980
- [Result] Di Felice V, Macaluso F, Montalbano A, Gammazza AM, Palumbo D, Angelone T, Bellafiore M, Farina F. Effects of conjugated linoleic acid and endurance training on peripheral blood and bone marrow of trained mice. J Strength Cond Res. 2007 Feb;21(1):193-8. doi: 10.1519/00124278-200702000-00035. PMID 17313269
- [Result] Diaz ML, Watkins BA, Li Y, Anderson RA, Campbell WW. Chromium picolinate and conjugated linoleic acid do not synergistically influence diet- and exercise-induced changes in body composition and health indexes in overweight women. J Nutr Biochem. 2008 Jan;19(1):61-8. doi: 10.1016/j.jnutbio.2007.01.006. Epub 2007 May 24. PMID 17531459
- [Result] Dilzer A, Park Y. Implication of conjugated linoleic acid (CLA) in human health. Crit Rev Food Sci Nutr. 2012;52(6):488-513. doi: 10.1080/10408398.2010.501409. PMID 22452730
- [Result] Eftekhari MH, Aliasghari F, Beigi MA, Hasanzadeh J. The effect of conjugated linoleic acids and omega-3 fatty acids supplementation on lipid profile in atherosclerosis. Adv Biomed Res. 2014 Jan 9;3:15. doi: 10.4103/2277-9175.124644. eCollection 2014. PMID 24600599
- [Result] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Result] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Result] Gaullier JM, Halse J, Hoivik HO, Hoye K, Syvertsen C, Nurminiemi M, Hassfeld C, Einerhand A, O'Shea M, Gudmundsen O. Six months supplementation with conjugated linoleic acid induces regional-specific fat mass decreases in overweight and obese. Br J Nutr. 2007 Mar;97(3):550-60. doi: 10.1017/S0007114507381324. PMID 17313718
- [Result] Hill AM, LaForgia J, Coates AM, Buckley JD, Howe PR. Estimating abdominal adipose tissue with DXA and anthropometry. Obesity (Silver Spring). 2007 Feb;15(2):504-10. doi: 10.1038/oby.2007.629. PMID 17299124
- [Result] Jenkins ND, Buckner SL, Cochrane KC, Bergstrom HC, Goldsmith JA, Weir JP, Housh TJ, Cramer JT. CLA supplementation and aerobic exercise lower blood triacylglycerol, but have no effect on peak oxygen uptake or cardiorespiratory fatigue thresholds. Lipids. 2014 Sep;49(9):871-80. doi: 10.1007/s11745-014-3929-0. Epub 2014 Jul 18. PMID 25034667
- [Result] Kennedy A, Martinez K, Schmidt S, Mandrup S, LaPoint K, McIntosh M. Antiobesity mechanisms of action of conjugated linoleic acid. J Nutr Biochem. 2010 Mar;21(3):171-9. doi: 10.1016/j.jnutbio.2009.08.003. Epub 2009 Dec 1. PMID 19954947
- [Result] Lambert EV, Goedecke JH, Bluett K, Heggie K, Claassen A, Rae DE, West S, Dugas J, Dugas L, Meltzeri S, Charlton K, Mohede I. Conjugated linoleic acid versus high-oleic acid sunflower oil: effects on energy metabolism, glucose tolerance, blood lipids, appetite and body composition in regularly exercising individuals. Br J Nutr. 2007 May;97(5):1001-11. doi: 10.1017/S0007114507172822. PMID 17381964
- [Result] Larsen TM, Toubro S, Astrup A. Efficacy and safety of dietary supplements containing CLA for the treatment of obesity: evidence from animal and human studies. J Lipid Res. 2003 Dec;44(12):2234-41. doi: 10.1194/jlr.R300011-JLR200. Epub 2003 Aug 16. PMID 12923219
- [Result] Mertz W, Tsui JC, Judd JT, Reiser S, Hallfrisch J, Morris ER, Steele PD, Lashley E. What are people really eating? The relation between energy intake derived from estimated diet records and intake determined to maintain body weight. Am J Clin Nutr. 1991 Aug;54(2):291-5. doi: 10.1093/ajcn/54.2.291. PMID 1858692
- [Result] Mitchell PL, Karakach TK, Currie DL, McLeod RS. t-10, c-12 CLA dietary supplementation inhibits atherosclerotic lesion development despite adverse cardiovascular and hepatic metabolic marker profiles. PLoS One. 2012;7(12):e52634. doi: 10.1371/journal.pone.0052634. Epub 2012 Dec 20. PMID 23285120
- [Result] Moon HS. Biological effects of conjugated linoleic acid on obesity-related cancers. Chem Biol Interact. 2014 Dec 5;224:189-95. doi: 10.1016/j.cbi.2014.11.006. Epub 2014 Nov 18. PMID 25446861
- [Result] Mougios V, Matsakas A, Petridou A, Ring S, Sagredos A, Melissopoulou A, Tsigilis N, Nikolaidis M. Effect of supplementation with conjugated linoleic acid on human serum lipids and body fat. J Nutr Biochem. 2001 Oct;12(10):585-594. doi: 10.1016/s0955-2863(01)00177-2. PMID 12031264
- [Result] Onakpoya IJ, Posadzki PP, Watson LK, Davies LA, Ernst E. The efficacy of long-term conjugated linoleic acid (CLA) supplementation on body composition in overweight and obese individuals: a systematic review and meta-analysis of randomized clinical trials. Eur J Nutr. 2012 Mar;51(2):127-34. doi: 10.1007/s00394-011-0253-9. Epub 2011 Oct 12. PMID 21990002
- [Result] Pariza MW, Park Y, Cook ME. Mechanisms of action of conjugated linoleic acid: evidence and speculation. Proc Soc Exp Biol Med. 2000 Jan;223(1):8-13. doi: 10.1046/j.1525-1373.2000.22302.x. PMID 10632956
- [Result] Pariza MW, Park Y, Cook ME. The biologically active isomers of conjugated linoleic acid. Prog Lipid Res. 2001 Jul;40(4):283-98. doi: 10.1016/s0163-7827(01)00008-x. PMID 11412893
- [Result] Pinkoski C, Chilibeck PD, Candow DG, Esliger D, Ewaschuk JB, Facci M, Farthing JP, Zello GA. The effects of conjugated linoleic acid supplementation during resistance training. Med Sci Sports Exerc. 2006 Feb;38(2):339-48. doi: 10.1249/01.mss.0000183860.42853.15. PMID 16531905
- [Result] Poirier P, Despres JP. Exercise in weight management of obesity. Cardiol Clin. 2001 Aug;19(3):459-70. doi: 10.1016/s0733-8651(05)70229-0. PMID 11570117
- [Result] Qi R, Yang F, Huang J, Peng H, Liu Y, Liu Z. Supplementation with conjugated linoeic acid decreases pig back fat deposition by inducing adipocyte apoptosis. BMC Vet Res. 2014 Jun 26;10:141. doi: 10.1186/1746-6148-10-141. PMID 24969229
- [Result] Riserus U, Arner P, Brismar K, Vessby B. Treatment with dietary trans10cis12 conjugated linoleic acid causes isomer-specific insulin resistance in obese men with the metabolic syndrome. Diabetes Care. 2002 Sep;25(9):1516-21. doi: 10.2337/diacare.25.9.1516. PMID 12196420
- [Result] Riserus U, Berglund L, Vessby B. Conjugated linoleic acid (CLA) reduced abdominal adipose tissue in obese middle-aged men with signs of the metabolic syndrome: a randomised controlled trial. Int J Obes Relat Metab Disord. 2001 Aug;25(8):1129-35. doi: 10.1038/sj.ijo.0801659. PMID 11477497
- [Result] Ritzenthaler KL, Shahin AM, Shultz TD, Dasgupta N, McGuire MA, McGuire MK. Dietary intake of c9,t11-conjugated linoleic acid correlates with its concentration in plasma lipid fractions of men but not women. J Nutr. 2012 Sep;142(9):1645-51. doi: 10.3945/jn.111.156794. Epub 2012 Jul 25. PMID 22833652
- [Result] Salas-Salvado J, Marquez-Sandoval F, Bullo M. Conjugated linoleic acid intake in humans: a systematic review focusing on its effect on body composition, glucose, and lipid metabolism. Crit Rev Food Sci Nutr. 2006;46(6):479-88. doi: 10.1080/10408390600723953. PMID 16864141
- [Result] Sluijs I, Plantinga Y, de Roos B, Mennen LI, Bots ML. Dietary supplementation with cis-9,trans-11 conjugated linoleic acid and aortic stiffness in overweight and obese adults. Am J Clin Nutr. 2010 Jan;91(1):175-83. doi: 10.3945/ajcn.2009.28192. Epub 2009 Nov 18. PMID 19923377
- [Result] Steck SE, Chalecki AM, Miller P, Conway J, Austin GL, Hardin JW, Albright CD, Thuillier P. Conjugated linoleic acid supplementation for twelve weeks increases lean body mass in obese humans. J Nutr. 2007 May;137(5):1188-93. doi: 10.1093/jn/137.5.1188. PMID 17449580
- [Result] Tarnopolsky M, Zimmer A, Paikin J, Safdar A, Aboud A, Pearce E, Roy B, Doherty T. Creatine monohydrate and conjugated linoleic acid improve strength and body composition following resistance exercise in older adults. PLoS One. 2007 Oct 3;2(10):e991. doi: 10.1371/journal.pone.0000991. PMID 17912368
- [Result] Thom E, Wadstein J, Gudmundsen O. Conjugated linoleic acid reduces body fat in healthy exercising humans. J Int Med Res. 2001 Sep-Oct;29(5):392-6. doi: 10.1177/147323000102900503. PMID 11725826
- [Result] Tsuboyama-Kasaoka N, Takahashi M, Tanemura K, Kim HJ, Tange T, Okuyama H, Kasai M, Ikemoto S, Ezaki O. Conjugated linoleic acid supplementation reduces adipose tissue by apoptosis and develops lipodystrophy in mice. Diabetes. 2000 Sep;49(9):1534-42. doi: 10.2337/diabetes.49.9.1534. PMID 10969838
- [Result] Wanders AJ, Brouwer IA, Siebelink E, Katan MB. Effect of a high intake of conjugated linoleic acid on lipoprotein levels in healthy human subjects. PLoS One. 2010 Feb 3;5(2):e9000. doi: 10.1371/journal.pone.0009000. PMID 20140250
- [Result] Zambell KL, Horn WF, Keim NL. Conjugated linoleic acid supplementation in humans: effects on fatty acid and glycerol kinetics. Lipids. 2001 Aug;36(8):767-72. doi: 10.1007/s11745-001-0783-8. PMID 11592726